CLINICAL TRIAL: NCT01662466
Title: A Randomized Double Blind Control Trial of Transdermal Testosterone Supplementation vs Placebo on Follicular Development and Atresia, Oocyte and Embryo Quality Among Women With Diminished Ovarian Reserve Undergoing in Vitro Fertilization
Brief Title: Effect of Testosterone Treatment on Embryo Quality
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Human Reproduction (Other)
Collaborators: Foundation for Reproductive Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 072312-01; CHR-DHEA-testosterone-2012 (Other: Center for Human Reproduction)
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-02

CONDITIONS: Primary Ovarian Insufficiency; Female Infertility Due to Diminished Ovarian Reserve
Keywords: testosterone; DHEA; IVF; egg quality; pregnancy rates
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Testosterone; Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA+Testosterone (Active Comparator): These patients will be administered the testosterone cream along with standard DHEA supplements
  Interventions: Drug: Testosterone cream (0.5mg per gram); Dietary Supplement: DHEA
- DHEA+Placebo (Placebo Comparator): These patients will receive the placebo cream along with her DHEA supplements. In other words, no testosterone will be administered.
  Interventions: Dietary Supplement: DHEA; Drug: Placebo

INTERVENTIONS:
Drug: Testosterone cream (0.5mg per gram) — Testosterone cream 2 gms per day applied transdermally to the left wrist to deliver 1.mg daily dose with estimated absorption of 100 ug per day testosterone
  Other Names: Testosterone
  Arms: DHEA+Testosterone
Dietary Supplement: DHEA — DHEA 25mg tid
  Other Names: Dehydroepiandrosterone
Drug: Placebo — Carrier cream without added testosterone in the identical type of pump
  Other Names: Carrier cream without added testosterone
  Arms: DHEA+Placebo

SUMMARY:
The purpose of this study is to determine the effect of treatment with trans-dermal testosterone cream compared to placebo on measures of ovarian reserve, oocyte and embryo quality, and pregnancy rates among women with evidence of diminished ovarian reserve that have persistently low serum testosterone and free testosterone after completing six previous weeks of DHEA supplementation.

DETAILED DESCRIPTION:
At CHR the investigators have been using DHEA supplementation to improve ovarian response to ovulation induction for in vitro fertilization for about five years (Barad, Brill et al. 2007; Barad, Weghofer et al .2009; Gleicher, Ryan et al. 2009; Gleicher, Weghofer et al. 2010; Gleicher and Barad 2011). Our views on the effect of androgens on the follicular environment have recently been reviewed (Gleicher, Weghofer et al. 2011). A recent analysis of androgen metabolites of DHEA in our patients suggested that women who successfully respond to DHEA supplementation with increased egg production and clinical pregnancy had testosterone above the normal median values for reproductive age women. There also appears to be a cohort of women who did not respond to DHEA and who had very low serum testosterone. The investigators decided to investigate if supplementing those women with testosterone to the normal female range would improve ovarian function and possibly increase pregnancy rates.

Recruitment & Experimental Plan

* A baseline blood draw following completion of 6 weeks of DHEA supplementation will determine eligibility for the study. The baseline blood determinations are part of the standard pre cycle screening at CHR for all patients.
* After signing informed consent subjects will be randomly assigned to either active testosterone cream treatment or placebo.
* Active treatment will consist of a testosterone delivery system that will deliver transdermal testosterone cream(0.5 mg per gram of cream.) The cream and placebo cream will be compounded by Metro Drugs (New York, NY) and dispensed in calibrated pump that will deliver one gram of cream per stroke. Transdermal absorption is about 10% so 2 grams (1.0 mg) per day applied to the skin will deliver about 100 ug per day. In preliminary analysis we have determined that a 2 gram dose of this preparation will raise total testosterone to our target range of between 50 and 100 ng/dL.
* The dose of testosterone cream will be 2 grams of cream per day applied to the left inner forearm. The study medication will continue to be applied for 6 weeks.
* All patients with evidence of diminished ovarian reserve in our practice are treated with DHEA. Thus, patients in this study will be receiving DHEA + testosterone or DHEA + Placebo. Patients who achieve a level of serum testosterone in the desired range using DHEA alone will not be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Women with 38 to 44 years old planning to undergo ovulation induction for IVF who are willing to sign an informed consent.
* BMI > 18 and <= 30 kg/m^2
* FSH > 10 mIU/mL
* AMH =< 1.05 ng/mL
* Using DHEA for treatment of DOR/POA.
* Baseline Total Testosterone less than 30 ng per deciliter (1.0 nmol per liter) or serum free testosterone concentrations of less than 3.5 pg per milliliter (12.1 pmol per liter), which are below the median values for normal premenopausal women (Endocrine Sciences, Calabasas Hills, Calif.).

Exclusion Criteria:

* History of hormone dependent neoplasm
* History of severe acne or hirsutism.
* Hyperlipidemia.
* Pre existing cardiac, renal or hepatic disease

Ages: 38 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-07-01; Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and Ongoing Pregnancy | 8 weeks post treatment initiation
  Clinical pregnancy is defined as the presence of a viable gestational sac visible in the uterus 4 weeks after embryo transfer. Clinical ongoing pregnancy is defined as intrauterine pregnancy with evidence of an active fetal heart at 6 weeks after embryo transfer.

SECONDARY OUTCOMES:
Measures of Atresia | 8 weeks after intervention initiation
  1. Follicular fluid will be collected separately for the first 5 follicles aspirated that are at least 18mm diameter for each patient.
  2. Granulosa cell counts will be performed on each follicle fluid. Granulosa cell counts of <10,000 per follicle will be considered atretic.
  3. Aliquots of follicular fluid will be analyzed for Testosterone, androstenedoine and estradiol using standard immuno assay. Healthy follicles should be capable of metabolizing testosterone to estradiol and should have a higher concentration estradiol (in nmol/ml) compared to testosterone
Oocytes number | 8 weeks after initiation of intervention
  The number of oocytes retrieved at oocyte retrieval for in-vitro fertilization will be compared between the treatment group and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Gleicher, MD, Study Chair — Center for Human Reproduction; David H Barad, MD, MS, Principal Investigator — Center for Human Reproduction
Locations (2):
- United States (2):
  - Center For Human Reproduction, New York, New York
  - Department of Medicine; Division of Endocrinology and Metabolism, University of Rochester School of Medicine and Dentistry, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- See also: Center For Human Reproduction Website — http://www.centerforhumanreprod.com/